CLINICAL TRIAL: NCT02545764
Title: The Effects of a Strength and Neuromuscular Exercise Programme for the Lower Extremity on Knee Load, Pain and Function in Obese Children and Adolescents: a Randomised, Single-blinded Controlled Trial
Brief Title: Training Induced Reduction of Lower-limb Joint Loads During Locomotion in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Pölten University of Applied Sciences (Other)
Collaborators: University of Vienna (Other); Medical University of Vienna (Other); Danube University Krems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LS13-009
Record Dates: First submitted 2015-08-28; First posted 2015-09-10 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Pediatric Obesity; Lower Extremity Biomechanics
Keywords: Gait Analysis; Knee Adduction Moment; Physiotherapy; Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Experimental): Strength and neuromuscular exercise programme
  Interventions: Other: Strength and neuromuscular exercise programme
- Control (No Intervention): Control group will receive opportunity for the training programme after data capturing is finished

INTERVENTIONS:
Other: Strength and neuromuscular exercise programme — 12 weeks strength and neuromuscular exercise programme for the lower extremity
  Arms: Intervention

SUMMARY:
Childhood obesity is one of the most critical and accelerating health challenges throughout the world. It is a major risk factor for developing varus/valgus misalignments of the knee joint. The combination of misalignment at the knee and excess body mass may result in increased joint stress and damage to articular cartilage. A training programme, which aims at developing a more neutral alignment of the trunk and lower limbs during movement tasks may be able to reduce knee loading during locomotion. Despite the large number of guidelines for muscle strength training and neuromuscular exercises that exists, most are not specifically designed to target the obese children and adolescent demographic.

The purpose of this study is to evaluate a training programme which combines strength and neuromuscular exercises specifically designed to the needs and limitations of obese children and adolescents and analyse the effects of the training programme from a biomechanical and clinical point of view.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 10 -18 years
* BMI greater than the 97th percentile
* Availability: can participate in two exercises session per week for a period of 12 weeks

Exclusion Criteria:

* Present syndromes
* Chronic joint diseases, osteoarthritic surgery or
* Neuro-motor diseases

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Overall peak external frontal knee moment and impulse | Baseline and 12 weeks
  Assessed by 3D gait analysis during walking

SECONDARY OUTCOMES:
Physical examination | Baseline and 12 weeks
  Changes of function and strength of the targeted muscle groups will be assessed by a physical therapist. Therefore, a hand-dynamometer to investigate differences in muscle strength will be used.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline and 12 weeks
  The Austria-German version of the Knee Injury and Osteoarthritis Outcome Score will be used to assess the participants' opinion about their knee.
Gait pattern | Baseline and 12 weeks
  Kinematics and external joint moments for the sagittal and frontal plane for hip, knee and ankle joints as well as spatio-temporal parameters will be assessed by 3D gait analysis during walking and stair climbing.
Adherence to the training programme | Participants will be followed for the duration of the intervention (12 weeks)
  Adherence will be considered as the percentage of actually completed sessions during the intervention period among the number of intended exercise sessions.
Ratings of knee related pain | Participants will be followed for the duration of the intervention (12 weeks)
  Ratings of knee related pain will be assessed using a 7-point ordinal scale.

OTHER OUTCOMES:
Cardiopulmonary testing | Baseline and 12 weeks
  The influence of the training programme on aerobic fitness will be assessed by submitting the participants to a symptom-limited cardiopulmonary exercise testing on a cycle ergometer.
Anthropometric measures | Baseline and 12 weeks
  The anthropometric evaluation will include the measurement of height, weight, waist circumference, hip circumference, waist-to-hip ratio and calculation of the body mass index.
Body Composition | Baseline and 12 weeks
  Body composition parameters will include, fat mass, fat free mass, total body water, body cell mass, extracellular mass and lean body mass.
Nutritional status | Baseline and 12 weeks
  The nutritional status will be assessed using the 24-hour recall method. This method records the daily, self-reported consumption of food-intake. In combination with a standardized nutritional food programme (EBISpro) the intake of macro- and micronutrients will be estimated.
Psychological status | Baseline and 12 weeks
  The AD-EVA test inventory as well as the Child Behavior Checklist (CBCL/4 -18 ) will be used to determine the psychological status of the participants.
Blood samples | Baseline and 12 weeks
  Quantification of routine blood sampling in obese patients and growth hormones and inflammation will be performed from venous blood samples in the Laboratory of the Department of Pediatrics and Adolescent Medicine at the Medical University of Vienna.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kreissl A, Jorda A, Truschner K, Skacel G, Greber-Platzer S. Clinically relevant body composition methods for obese pediatric patients. BMC Pediatr. 2019 Mar 21;19(1):84. doi: 10.1186/s12887-019-1454-2. PMID 30898093
- [Derived] Horsak B, Schwab C, Baca A, Greber-Platzer S, Kreissl A, Nehrer S, Keilani M, Crevenna R, Kranzl A, Wondrasch B. Effects of a lower extremity exercise program on gait biomechanics and clinical outcomes in children and adolescents with obesity: A randomized controlled trial. Gait Posture. 2019 May;70:122-129. doi: 10.1016/j.gaitpost.2019.02.032. Epub 2019 Feb 27. PMID 30851623
- [Derived] Horsak B, Artner D, Baca A, Pobatschnig B, Greber-Platzer S, Nehrer S, Wondrasch B. The effects of a strength and neuromuscular exercise programme for the lower extremity on knee load, pain and function in obese children and adolescents: study protocol for a randomised controlled trial. Trials. 2015 Dec 23;16:586. doi: 10.1186/s13063-015-1091-5. PMID 26700568